CLINICAL TRIAL: NCT01893112
Title: Reducing HIV Stigma to Improve Health Outcomes for African-American Women
Brief Title: Reducing HIV Stigma for African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Alabama at Birmingham (Other); Northwestern University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Deepa Rao, Associate Professor, Department of Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 43970; R01MH098675 (NIH)
Record Dates: First submitted 2013-02-11; First posted 2013-07-08 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Unity Workshop (Experimental): The intervention is a workshop facilitated by a peer advocate (an African American woman who is also HIV positive) and a social worker. It has exercises, videos and group discussions intended to equip participants with coping skills to overcome HIV related stigma and the negative outcomes related to stigma. The workshop will last about 8 hours total across 2 two days (4 hours per day). The researcher in the current study has done a lot of work in adapting this intervention for African American women. The workshop has been piloted in Seattle and had promising results. Based on results in the pilot study, a 2 hour booster session has been added 6 months after the initial workshop
  Interventions: Behavioral: Unity Workshop
- Breast Cancer Screening (Other): The time and attention control group workshop will be facilitated by a research coordinator. The control group program is based on another program that is designed explore issues related to breast cancer screening among African American women. The program has the same format as the Unity Workshop, with video and group discussion. Although breast cancer may be associated with stigma, we anticipated that breast cancer stigmas would not be related to HIV-associated stigma, which is our primary outcome of interest. The control groups will be held during the same week as the Unity Workshops, and control group participants will complete assessments on the same schedule as the Unity Workshop participants.
  Interventions: Behavioral: Breast Cancer Screening

INTERVENTIONS:
Behavioral: Unity Workshop — The intervention is based on other stigma reduction programs that are being used internationally (HIV Stigma Toolkit developed by the International Center for Research on Women and trigger videos developed by International Training & Education Center for health).
  Arms: Unity Workshop
Behavioral: Breast Cancer Screening
  Arms: Breast Cancer Screening

SUMMARY:
African American women account for 66% of HIV infections in women in the U.S., AIDS is a leading cause of death for African American women, and African Americans have the lowest medication adherence rates compared to other groups in the U.S. One of the reasons for low medication adherence among African Americans is fear of stigma. HIV stigma has been linked to depression, psychological distress, poor quality of life, poor medication adherence and service utilization contributing to morbidity and mortality. Research has found that stigma is a moderator to poor adherence via depressive symptoms.

The current study is a randomized control trial with a time and attention control group to test the effectiveness of a stigma reduction intervention adapted for use with African American women. A total of 224 African American women will be recruited to participate in the study. Half of the women will be from Chicago, Illinois (112) and the other half will be from Birmingham, Alabama (112). A workshop will be held once a study site has recruited 28 women, half of the women will be in the intervention group (14) and the other half will be in the control group (14). Each study site will have 4 cohorts of 28 women.

The main aims of the current study are:

1. to determine the long-term effectiveness of the intervention to reduce stigma for African American women living with HIV in Chicago Illinois and Birmingham, Alabama
2. to examine whether stigma reduction due to the intervention is associated with improved physical health biomarkers (CD4+ T cell count, viral load), mediated by reduced psychological symptoms (depressive symptoms), improved engagement to care, and improved medication adherence
3. to explore whether stigma reduction due to the intervention is moderated by location (Chicago vs. Birmingham), transmission risk factor, time since diagnosis, and perceived social support

We expect that the multimedia workshop intervention will demonstrate effectiveness in reducing internalized stigma through an easily-disseminated method, and that it will have a positive impact on medication adherence and engagement in care for African American women living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* they are women who identify as having an African American racial/ethnic background
* born in the U.S. (including women of Caribbean origin if born in the U.S.
* speak and understand English as their primary language of communication outside the home
* they are 18 years of age or older
* have a documented HIV positive status (women are on antiretroviral treatment and women who are not on antiretroviral are eligible)
* able to see and interact with a touchscreen computer in English.

Exclusion Criteria:

* women who not self-identify as African American
* women who are African born or born outside the United States
* younger than 18 years of age
* unable to provide informed consent
* life expectancy less than 1 year per physician report
* unable to see and interact with a touchscreen computer in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-06; Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in stigma scores from baseline to 12 months. | baseline, after intervervention, 4 months, 6 months, 8 months, 12 months
  We will see if the intervention/workshop reduces HIV related stigma after 1 year in the study. We will use the Stigma Scale for Chronic Illness to measure stigma.

SECONDARY OUTCOMES:
Location as a moderator variable | baseline, after intervervention, 4 months, 6 months, 8 months, 12 months
  This is a multi-site study (Chicago and Birmingham) and we are interested in seeing if location is a moderating variable
Post-Traumatic Stress Disorder Checklist | baseline, 12 months
Adherence to HIV Medication | baseline, after intervention, 4 months, 6 months, 8 months, 12 months
  Adherence to HIV medication will be measured by participants self report of adherence using commonly used set of questions.
Patient Health Questionnaire (PHQ-9) | baseline, after intervention, 4 months, 6 months, 8 months, 12 months
  We will look at the correlation between stigma scores and depression scores over time.
Medical Outcomes Study Social Support Scale | Study duration
  We are going to use a validated social support scale, and analyze social support as a correlate.
substance abuse | baseline, 12 months
  substance use and stigma of substance use will be measured using: Alcohol Use disorders Identification Test (AUDIT) Severity of Dependence Scale (SDS) Substance Abuse Self Stigma (SASS)
Engagement in Care (from patient record) | baseline, 4 months, 8 months, 12 months
  Research assistants will access participants' medical records to see if patients have missed any HIV related visits (i.e. medical, counseling). Engagement to care will be measured as a proportion (missed visits over total scheduled). Rescheduled visits will not count as missed visits. At baseline, we will look at visits for the past 12 months.
HIV viral load (from medical chart) over 1 year study duration | baseline, 4 months, 8 months, 12 months
  We want to examine whether stigma reduction due to the intervention is associated with improved physical health bio-markers such as suppression in HIV viral load in the blood (taken from medical chart/previous clinical blood tests).
Change in CD4 count | baseline, 4 months, 8 months, 12 months
  We want to see wither stigma reduction from the intervention associated with improved physical health bio-markers such as CD4+ T cell count.

CONTACTS AND LOCATIONS:
Overall Officials: Deepa Rao, PhD, MA, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Northwestern University (NU), Chicago, Illinois

REFERENCES:
- [Background] CDC. HIV/AIDS Surveillance Report: Cases of HIV infection and AIDS in the United States. 2004.
- [Background] CDC. Web-based Injury Statistics Query and Reporting System (WISQARS) [online]. Leading Cause of Death for Black Women 1999-2007. 2008; www.cdc.gov/ncipc/wisqars. Accessed December 4, 2011.
- [Background] Halkitis PN, Parsons JT, Wolitski RJ, Remien RH. Characteristics of HIV antiretroviral treatments, access and adherence in an ethnically diverse sample of men who have sex with men. AIDS Care. 2003 Feb;15(1):89-102. doi: 10.1080/095401221000039798. PMID 12655837
- [Background] Palacio H, Kahn JG, Richards TA, Morin SF. Effect of race and/or ethnicity in use of antiretrovirals and prophylaxis for opportunistic infection: a review of the literature. Public Health Rep. 2002 May-Jun;117(3):233-51; discussion 231-2. doi: 10.1093/phr/117.3.233. PMID 12432135
- [Background] Traeger L, O'Cleirigh C, Skeer MR, Mayer KH, Safren SA. Risk factors for missed HIV primary care visits among men who have sex with men. J Behav Med. 2012 Oct;35(5):548-56. doi: 10.1007/s10865-011-9383-z. Epub 2011 Nov 9. PMID 22068878
- [Background] Rao D, Kekwaletswe TC, Hosek S, Martinez J, Rodriguez F. Stigma and social barriers to medication adherence with urban youth living with HIV. AIDS Care. 2007 Jan;19(1):28-33. doi: 10.1080/09540120600652303. PMID 17129855
- [Background] Rintamaki LS, Davis TC, Skripkauskas S, Bennett CL, Wolf MS. Social stigma concerns and HIV medication adherence. AIDS Patient Care STDS. 2006 May;20(5):359-68. doi: 10.1089/apc.2006.20.359. PMID 16706710
- [Background] Rao D, Feldman BJ, Fredericksen RJ, Crane PK, Simoni JM, Kitahata MM, Crane HM. A structural equation model of HIV-related stigma, depressive symptoms, and medication adherence. AIDS Behav. 2012 Apr;16(3):711-6. doi: 10.1007/s10461-011-9915-0. PMID 21380495
- [Background] Rao D, Desmond M, Andrasik M, Rasberry T, Lambert N, Cohn SE, Simoni J. Feasibility, acceptability, and preliminary efficacy of the unity workshop: an internalized stigma reduction intervention for African American women living with HIV. AIDS Patient Care STDS. 2012 Oct;26(10):614-20. doi: 10.1089/apc.2012.0106. Epub 2012 Sep 17. PMID 22984780